CLINICAL TRIAL: NCT05284253
Title: Is There an Allergy to Pure Metallic Gold Microparticles?: A Epicutaneous Test of Gold Microparticles, Gold Thiosulphate and Placebo.
Brief Title: Is There an Allergy to Pure Metallic Gold Microparticles?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Sten Rasmussen, MD, PhD, Professor Head of Department of Clinical Medicine, Aalborg University
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NorthernODD
Record Dates: First submitted 2021-11-21; First posted 2022-03-17 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Allergic Reaction
MeSH Terms: conditions — Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold microparticles (Experimental): Metallic gold microparticles, 20-micron diameter, 1 % w/v in petrolatum
  Interventions: Other: Gold microparticles
- Gold thiosulphate (Active Comparator): Gold Sodium Thio Sulphate, 1 % w/v in petrolatum
  Interventions: Other: Gold thiosulphate

INTERVENTIONS:
Other: Gold microparticles — Metallic gold microparticles, 20-micron diameter, 1 % w/v in petrolatum
  Other Names: Patch test
  Arms: Gold microparticles
Other: Gold thiosulphate — Gold Sodium Thio Sulphate, 1 % w/v in petrolatum
  Other Names: Patch test
  Arms: Gold thiosulphate

SUMMARY:
The investigators hypothesize gold is inert and thereby there is no pure-gold allergy. The primary aim of this study is to measure the prevalence of allergy to metallic pure gold microparticles and allergy to GSTS.

DETAILED DESCRIPTION:
TRUE test panel which includes gold sodium thiosulphate (GSTS), 1 % w/v in petrolatum, and gold microparticles, 20-micron diameter, 1 % w/v in petrolatum, will be added added to the baseline series. It will be applied to the upper back of healthy adults in aluminum Finn Chamber for 48 hours. Clinical evaluation will be performed 24 hours after removal the test according to standard procedures for evaluation of epi-cutaneous challenging (Johansen 2015).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic dermatitis

Exclusion Criteria:

* age < 18

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Patch test | 72 hours
  Test materials will be applied on the upper back of the volunteers in aluminium Finn Chambers for 48 hours. Clinical evaluation will be performed 24 hours after removal of the test substances according to standard procedures for evaluation of epicutaneous challenging according to criteria of ICDRG (International Contact Dermatitis Research Group) (Johansen 2015). Reactions: doubtfull, faint macular erythema only; weak positive reaction, erythema, infiltration papules; strong positive reaction, erythema, infiltration, papular, vesicles; erythema positive reaction, intense erythema, infiltration and coalescing vesicles; negative reaction; irritant reaction; not tested

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, PhD, Principal Investigator — Department of Clinical Medicine, Aalborg Unviversity

IPD SHARING:
Plan to Share IPD: Undecided